CLINICAL TRIAL: NCT02591875
Title: Atrial Flutter Ablation in a Real World Population: A Multicenter Italian Registry (The LEONARDO Study)
Brief Title: Atrial Flutter Ablation in a Real World Population
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Azienda Ospedaliera Pugliese Ciaccio (Other)
Responsible Party: Principal Investigator, Giampiero Maglia, Head of Electrophysiology and Cardiac Pacing, Azienda Ospedaliera Pugliese Ciaccio
Other Study IDs: Protocollo n. 156 (06/11/2015)
Record Dates: First submitted 2015-10-07; First posted 2015-10-30 (Estimated); Last update posted 2016-10-19 (Estimated); Status verified 2016-10

CONDITIONS: Atrial Flutter
Keywords: Cardiac Catheter Ablation; Cardiac Arrhythmias; Atrial Flutter
MeSH Terms: conditions — Atrial Flutter; Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The "LEONARDO" study is a non-randomized, multicenter, prospective study in which consecutive patients indicated for Atrial Flutter isthmus-dependent (AFL) ablation will be enrolled. Patients can be treated with any market released catheter for ablation. The decision to perform the ablation of AFL will be made based on clinical evaluation of the investigators according to their clinical practice. The study does not require specific surgical techniques. Patient time commitment for the study is approximately 12 months.The study has been designed to describe the italian clinical practice in relation to the approach of AFL ablation. In particular, the investigators will describe the methods for the validation of ablation success, the techniques adopted, and the patient management approaches in the participating centers.

DETAILED DESCRIPTION:
Catheter ablation of Atrial Flutter has become an accepted alternative to pharmacologic therapy.The current guidelines recommend the catheter ablation at the first episode of AFL (Class IIa) or in any case of recurrent episodes of AFL (Class I). Recent studies have already demonstrated a high degree of procedural efficacy (higher than 90%). However, there are still two main areas of investigation. First, what is the best method to obtain an effective lesion. Second, what is the most reliable method to validate the procedure success.The present study is aimed at investigating these aspects in the current Italian clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Patient undergoing ablation of atrial flutter isthmus-dependent
* Patient able to sign an authorization to use and disclose health information or an Informed Consent.
* Patient available to attend scheduled follow-up visits at the center for at least 12 months

Exclusion Criteria:

* Patient is participating in another clinical study that may have an impact on the study endpoints

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All consecutive patients, clinically indicated for an atrial flutter ablation, will be enrolled after signing of an informed consent form and an authorization to use and disclose health information.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2015-10; Primary Completion 2020-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of Subjects With Complete Bidirectional Conduction Block | Time Frame: within 30 minutes after ablation procedure
  Acute success is defined as the confirmation of complete bidirectional conduction block across the cavo-tricuspid isthmus. The percentage of subjects with confirmed conduction block will serve as the outcome measure.

SECONDARY OUTCOMES:
Recurrence of symptoms of AFL, measured as the proportion of patients reporting symptoms during follow-up | 12 months
  number of patients with symptoms of AFL during follow-up
Recurrence of AFL, measured as the proportion of patients with an episode longer than 30s documented at 24h Holter ECG recording during follow-up | 12 months
  number of patients with recurrence of AFL documented at ECG recording during follow-up
Lesion's validation criteria | an average of 12 months following the ablation procedure
  agreement between acute ablation success and long-term absence of AFL recurrence
Ablation procedure time | intraoperative
  * RadioFrequency time;
  * ablation time;
  * Fluoroscopy time
Acute adverse events | intraoperative
Adverse Events during Follow up | 12 months

CONTACTS AND LOCATIONS:
Locations (4):
- Italy (4):
  - Clinica Montevergine, Mercogliano, AV
  - Fondazione Poliambulanza - Istituto Ospedaliero, Brescia, BS
  - Presidio Ospedaliero Policlinico Casilino, Roma, RM
  - Azienda Ospedaliera Pugliese-Ciaccio, Catanzaro

REFERENCES:
- [Derived] Maglia G, Pentimalli F, Verlato R, Solimene F, Malacrida M, Aspromonte V, Bacino L, Turrini P, Infusino T, La Greca C, Perego GB, Papa AA, De Ruvo E, Zingarini G, Devecchi C, Scaglione M, Tomasi C, Pirrotta S, Stabile G. Ablation of CTI-dependent flutter using different ablation technologies: acute and long-term outcome from the LEONARDO study. J Interv Card Electrophysiol. 2023 Oct;66(7):1749-1757. doi: 10.1007/s10840-023-01519-7. Epub 2023 Mar 4. PMID 36869990